CLINICAL TRIAL: NCT00801827
Title: PET Imaging and Bariatric Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Julia P.Dunn,MD, Physician, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB#061246
Record Dates: First submitted 2008-12-02; First posted 2008-12-04 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-01

CONDITIONS: Obesity, Morbid
Keywords: Obesity; Addiction; PET imaging
MeSH Terms: conditions — Obesity, Morbid; Obesity; Behavior, Addictive | interventions — fallypride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- F-18 (fallypride) (Experimental): Subjects undergoing bariatric surgery will have Positron Emission Tomography (PET) scans of their brains using F-18 (fallypride), a dopamine type 2/3 (DA D2/3) receptor radioligand whose binding is sensitive to competition with endogenous dopamine, before and after the operation.
  Interventions: Drug: F-18 (fallypride)

INTERVENTIONS:
Drug: F-18 (fallypride) — Subjects undergoing bariatric surgery will have Positron Emission Tomography (PET)scans of their brains using the radioligand fallypride before and after the operation.

SUMMARY:
The purpose of this study is to look at certain areas of the brain that are related to addictive behaviors, such as overeating. These areas are called 'dopamine type 2 receptors' (DRD2/3) and other studies have shown that obese people have less of these. We propose that low DRD2/3 availability seen in morbidly obese subjects will change with weight loss associated with bariatric surgery.

DETAILED DESCRIPTION:
The purpose of this study is to look at certain areas of the brain that are related to addictive behaviors, such as overeating. These areas are called 'dopamine type 2 receptors' (DRD2/3) and other studies have shown that obese people have less of these. We propose that low DRD2/3 availability seen in morbidly obese subjects will change with weight loss associated with bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-60 years
* BMI equal to or greater than 40, or equal to or greater than 35 if there are 2 or more co-morbidities
* Weight less than 350 pounds

Exclusion Criteria:

* History of substance abuse,including but not limited to alcohol, cocaine, marijuana, heroin, nicotine
* History of psychiatric disorders
* Use of any antidepressants or psychotropics in the past 12 months
* Diabetes Mellitis
* Positive pregnancy test
* Any condition felt by the PI or co-investigators to interfere with the individual's ability to complete the study
* Subjects on medications for the last 3 months, such as sibutramine, which could affect the quality of the study, as determined by the PI
* Inability to travel to Nashville, TN four times

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2007-01; Primary Completion 2011-03 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia P Dunn, MD, Principal Investigator — Vanderbilt University Medical Center; Robert M Kessler, MD, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 patients consented to the study but 2 never participated due to scheduling conflicts. All 5 participants that started the study went on to complete the study.
Groups:
- Surgical: Patients approved for RYGB or VSG surgery for weight loss at Vanderbilt University Medical Center were recruited.
Period: Overall Study
Arm/Group | Surgical
Started | 5 (2 others consented but due to scheduling did not complete)
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Surgical
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (4.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Preop BMI [Mean (Standard Deviation); unit: kg/m^2] | 43.2 (6.26)

OUTCOME MEASURES:

1. Primary Outcome: Regional DRD2/3 Binding Percent Changes After Bariatric Surgery
Time Frame: ~7 weeks
Measure: Mean (Standard Deviation); unit: percentage of binding potential change
Groups:
- F-18 (Fallypride): Subjects undergoing bariatric surgery will have Positron Emission Tomography (PET) scans of their brains using F-18 (fallypride), a dopamine type 2 (DA D2) receptor radioligand whose binding is sensitive to competition with endogenous dopamine, before and after the operation.
Arm/Group | F-18 (Fallypride)
Number analyzed (Participants) | 5
percentage of binding potential change
  Caudate | -10.14 (2.74)
  Putamen | -9.39 (6.67)
  Ventral Striatum | -8.11 (3.90)
  Hypothalamus | -8.76 (2.52)
  Substania nigra | -10.2 (1.78)
  Medial thalamus | -8.17 (2.10)
  Amygdala | -8.99 (2.52)

ADVERSE EVENTS:
Arm/Group | F-18 (Fallypride)
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes